CLINICAL TRIAL: NCT06548568
Title: A Two-year Non-interventional, Real-world, Observational Study to Assess Safety of OZURDEX® (Dexamethasone Intravitreal Implant) in Patients With Diabetic Macular Edema in China
Brief Title: A Real-world Study to Assess Safety of OZURDEX® (Dexamethasone Intravitreal Implant) in Adult Participants With Diabetic Macular Edema in China
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-425
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; OZURDEX

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OZURDEX: Participants with diabetic macular edema prescribed OZURDEX in routine clinical practice are observed from the first dose for up to 24 months.

SUMMARY:
The dexamethasone intravitreal implant (OZURDEX) delivers dexamethasone gradually to the retina over time. It is an approved drug for the treatment of diabetic macular edema (DME). This study will assess the long-term safety and effectiveness of OZURDEX in adult participants with DME in the routine clinical setting in China.

Approximately 110 participants who are prescribed OZURDEX by their physicians will be enrolled in multiple medical institutions in China where OZURDEX is used for DME in routine clinical practice.

Participants will be followed for 24 months after the first administration of OZURDEX according to the routine clinical practice of the prescribing centers. A subsequent 30-day follow-up after the last dose will be performed to obtain information on any new or ongoing safety events and concomitant medications.

No additional burden for participants in this trial is expected.

ELIGIBILITY:
Inclusion Criteria:

- Participant scheduled to receive at least one intravitreal OZURDEX® injection for DME as per most current local approved label after its approval for DME in China.

Exclusion Criteria:

* Concurrent participation in interventional clinical research that required treatment or use of an investigational agent.
* Participants for whom OZURDEX® is contraindicated:

  * Participants with known hypersensitivity to OZURDEX® or any components of this product.
  * Participants with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
  * Participants with late stage glaucoma that cannot be controlled with medication alone.
  * Aphakia with ruptured posterior lens capsule.
  * Eyes with anterior chamber intraocular lenses (ACIOL), iris- or scleral-fixated intraocular lenses, and ruptured posterior lens capsule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample: participants with diabetic macular edema (DME) who resided in China.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs), including Adverse Events of Special Interest (AESIs) | Up to approximately 24 months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The AESIs can include the following: cataracts, elevated IOP and conjunctival hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- China (13):
  - Peking University People'S Hospital /ID# 274505, Beijing, Beijing Municipality
  - Xiamen Eye Center of Xiamen University /ID# 268172, Xiamen, Fujian
  - Zhongshan Ophthalmic Center,SunYat-Sen University /ID# 274555, Guangzhou, Guangdong
  - Henan Provincial Eye Hosptial /ID# 272424, Zhengzhou, Henan
  - General Hospital of Central Theater Command /ID# 273618, Wuhan, Hubei
  - The First Affiliated Hospital of Dalian Medical University /ID# 270563, Dalian, Liaoning
  - Xi'an Fourth Hospital /ID# 270562, Xi'an, Shaanxi
  - Qingdao Eye Hospital Of Shandong First Medical University /ID# 268173, Qingdao, Shandong
  - Shanghai General hospital /ID# 270376, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University /ID# 273656, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 273617, Hangzhou, Zhejiang
  - The Affiliated Eye Hospital Of Wenzhou Medical University /ID# 274466, Wenzhou, Zhejiang
  - Shanxi Eye Hospital /ID# 270564, Taiyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-425